CLINICAL TRIAL: NCT05931692
Title: The Role of Virtual Reality in Examining the Effect of Fear of Falling (FOF) on Postural Stability in Individuals Without and With Parkinson's Disease in Egypt: A Mixed Methods Feasibility Study
Brief Title: Virtual Reality and Fear of Falling in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: Ahram Canadian University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasmine Gomaa, Lecturer of Physcial Therapy for Neuromuscular Disorders, Ahram Canadian University
Other Study IDs: P.T/ NEUR /3/2023/46
Record Dates: First submitted 2023-06-15; First posted 2023-07-05 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Parkinson; Parkinson Disease; Parkinson's Disease and Parkinsonism
MeSH Terms: conditions — Parkinson Disease; Parkinsonian Disorders | interventions — Exergaming; Electroencephalography; Electromyography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals without Parkinson's disease: People over 40 years old
  Interventions: Diagnostic Test: Virtual reality; Diagnostic Test: Electroencephalogram; Diagnostic Test: Electromyography; Diagnostic Test: Motion Capture system; Diagnostic Test: Polar H10 Heart Sensor; Diagnostic Test: Inertial measurement Unite
- Parkinson Disease: People over 40 years old who have Parkinson's Disease at stage I to III Hoehn and Yahr scale
  Interventions: Diagnostic Test: Virtual reality; Diagnostic Test: Electroencephalogram; Diagnostic Test: Electromyography; Diagnostic Test: Motion Capture system; Diagnostic Test: Polar H10 Heart Sensor; Diagnostic Test: Inertial measurement Unite

INTERVENTIONS:
Diagnostic Test: Virtual reality — Virtual environment that triggers fear of falling
Diagnostic Test: Electroencephalogram — Detect brain waves in response to fear of falling
Diagnostic Test: Electromyography — Measures muscle activity and response to fear of falling
Diagnostic Test: Motion Capture system — Measures postural and gait responses to fear of falling
Diagnostic Test: Polar H10 Heart Sensor — Heart rate monitor
Diagnostic Test: Inertial measurement Unite — Measure Postural sway

SUMMARY:
Background: Falls are common in elderly individuals and those with neurological conditions like Parkinson's disease. Parkinson's disease causes postural instability and mobility issues that lead to falls and reduced quality of life. The fear of falling (FoF), a natural response to unstable balance, can exacerbate postural control problems. However, evaluating FoF relies primarily on subjective self-reports due to a lack of objective assessment methods.

Objectives: This mixed-methods feasibility study aims to develop an objective method for assessing fear of falling during motion and walking using virtual reality. This protocol examines a range of FoF-related responses, including cognitive, neuromuscular, and postural stability factors.

Methods: Individuals without and with Parkinson's disease will complete questionnaires, movement tasks, and walking assessments in real and virtual environments where FoF can be elicited using virtual reality (VR) technology. Data from center-of-pressure measurements, electromyography, heart rate monitoring, motion capture, and usability metrics will evaluate the method's acceptability and safety. Semi-structured interviews will gather participants' and researchers' experiences of the protocol.

Discussion: This method may allow accurate assessment of how FoF impacts movement by measuring cognitive, neuromuscular, and postural responses during gait and motion. Virtual environments reproduce real-life scenarios that trigger FoF. Rigorously assessing FoF with this approach could demonstrate its ability to quantify the effects of FoF on movement.

Conclusions: This protocol aims to improve FoF assessment by evaluating multiple responses during movement in virtual environments. It addresses current measures' limitations. A feasibility study will identify areas for improvement specific to Parkinson's disease. Successful validation could transform how FoF is evaluated and managed.

ELIGIBILITY:
Inclusion Criteria:

* People ≥ 40 years old.
* Participants diagnosed with Parkinson's disease by a neurologist, regardless the type.
* Modified Hoehn and Yahr stages I to III.
* Able to follow instructions and understand questions.
* Able to walk independently and without walking aids.
* People who experience excessive fear of falling and fear of movement.
* Able to communicate verbally.
* Stable use of Parkinson's Disease or other comorbidities medications.

Exclusion Criteria:

* Impaired vision and hearing.
* Unstable medical condition.
* Co-existing neurological or orthopedic conditions that may limit mobility and affect participation.
* Dizziness, vertigo, headache, and motion-sickness.
* Cognition impairments.
* Pregnancy.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two groups of participants, who age 40 or older, will be involved in this study. Each group will have from 10 to 30 participants. The first group will include a group of individuals without Parkinson's disease and the second group will include people with Parkinson's disease, both will be screened for eligibility. Participants who meet the inclusion criteria will go through the planned assessment procedure.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-07-17 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Movement Control | 5 minutes
  Movement control throughout the movement scenario will be assessed using a Qualisys motion capture system (MCS).
Balance Assessment | 5 minutes
  Force platforms will measure the center of pressure (COP) displacement during the movement scenario.
Postural Sway | 5 minutes
  A postural Inertial Measurement Unit (IMU) will be placed over the projected center of mass located at the 4th lumbar vertebra to evaluate postural sway.
EEG Monitoring | 5 minutes
  The electroencephalogram (EEG) will be used to monitor the neuromuscular system's reaction to fear throughout the movement scenario. power in alpha and beta frequency bands will be recorded.
EMG Monitoring | 5 minutes
  The electromyography (EMG) will be employed to monitor the neuromuscular system's reaction to fear throughout the movement scenario. Muscle activation of lower limb muscles such as tibialis anterior and quadriceps will be recorded by surface EMG.
Heart Rate Monitoring | 5 minutes
  The unit of measurement for heart rate monitoring is typically beats per minute (BPM). The Polar H10 heart rate sensor will be used in to measure the electrical signals produced by the heart and provides continuous and accurate heart rate readings in BPM.
Suitability Evaluation | 30 minutes
  the Suitability Evaluation Questionnaire (SEQ) is the SEQ Suitability Evaluation Questionnaire for Virtual Rehabilitation Systems. The range of scores is 0 to 100, with higher scores indicating a better outcome. The SEQ is scored by summing the responses to the 14 items. The items are scored on a 7-point Likert scale, with 1 = strongly disagree and 7 = strongly agree. The total score can range from 0 to 98. A higher score on the SEQ indicates that the VR system is perceived as being more user-friendly, enjoyable, and safe. This suggests that the patient is more likely to use the VR system and to benefit from it.
Sense of Presence | 30 minutes
  The iGroup Presence Questionnaire (IPQ) has a range of scores is 0 to 6, with higher scores indicating a better outcome. The IPQ is scored by summing the responses to the 14 items. The items are scored on a 7-point Likert scale, with 1 = disagree strongly and 7 = agree strongly. The total score can range from 0 to 98. A higher score on the IPQ indicates that the user feels more present in the Virtual environment (VE). This suggests that the VE is more immersive and engaging, and that the user is more likely to be absorbed in the experience.
Effort | 30 minutes
  The Borg Rated Perceived Exertion (RPE) scale will record effort during the session. The Borg Rated Perceived Exertion (RPE) Scale: Range 0-10, higher scores indicate greater perceived exertion.
Adverse events | 30 minutes
  any adverse events during the procedure and after effects will be documented. Number of participants reporting adverse events as per study protocol

SECONDARY OUTCOMES:
Fear of Falling Assessment | 45 minutes
  Fear of falling will be assessed using the Falls Efficacy Scale International (FES-I).
Cognition Assessment | 45 minutes
  Montreal Cognitive Assessment (MoCA) is a brief, 30-item cognitive screening test that is used to assess a person's cognitive abilities. Montreal Cognitive Assessment has a minimum value of 0 and maximum value of 3 with Higher score indicates better outcome. A score of 26 or higher is considered normal, while a score of 25 or lower may indicate cognitive impairment.
Depression Assessment | 45 minutes
  Hamilton Depression Rating Scale (HAM-D) will be used to assess depression level. Minimum value is 0 and the maximum value is 52. Lower scores indicate better outcome. The HAM-D is a 17-item clinician-rated scale that is used to assess the severity of depression. The scale was developed by Max Hamilton in 1960 and has been used in a wide range of studies to assess depression. The HAM-D covers a range of symptoms of depression, including depressed mood, feelings of guilt, suicidal ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. Each item is scored on a 5-point scale, with 0 = absent and 4 = severe. The total score can range from 0 to 52, with a higher score indicating more severe depression.
Anxiety Assessment | 45 minutes
  Hamilton Anxiety Rating Scale will be used to assess level of anxiety. the Minimum value is 0 and Maximum value is 56. Lower score indicates better outcome. It is a 14-item clinician-rated scale that is used to assess the severity of anxiety. The scale was developed by Max Hamilton in 1959 and has been used in a wide range of studies to assess anxiety. It covers a range of symptoms of anxiety, including anxious mood, tension, fears, insomnia, intellectual, somatic (muscular), somatic (sensory), cardiovascular, respiratory, gastrointestinal, genitourinary, autonomic symptoms, and behavior at interview. Each item is scored on a 4-point scale, with 0 = absent and 4 = severe. The total score can range from 0 to 56, with a higher score indicating more severe anxiety.
Participation Assessment | 45 minutes
  Participation levels will be assessed using the World Health Organization Disability Assessment Schedule 2.0. the Minimum value is 0 and Maximum value is 100. Lower score indicates better outcome. The WHODAS 2.0 is a 12-item self-report questionnaire that is used to assess the impact of a health condition on an individual's functioning. The items are scored on a 5-point scale, with 0 = no difficulty and 4 = extreme difficulty. The total score can range from 0 to 100, with a lower score indicating less disability. The WHODAS 2.0 covers six domains of functioning: cognition, mobility, self-care, getting along, life activities, and participation. The scale was developed by the World Health Organization (WHO) and is based on the International Classification of Functioning, Disability and Health (ICF).
Health-related Quality of Life Assessment | 45 minutes
  Health-related quality of life will be evaluated using the Parkinson's Disease Questionnaire 39 (PDQ-39). Parkinson's Disease Questionnaire 39 has a Minimum value of 0 and Maximum value of 100. Lower score indicates better outcome. The PDQ-39 is a 39-item self-report questionnaire that is used to assess the impact of Parkinson's disease (PD) on an individual's quality of life. The items are scored on a 5-point scale, with 0 = no problem and 4 = severe problem. The total score can range from 0 to 100, with a lower score indicating better quality of life.
Balance confidence | 10 minutes
  Balance confidence will be evaluated using Activity-specific Balance Confidence scale (ABC scale). Which is a self-administered scale to indicate the level of confidence the person has in doing the activity without losing his/her balance. The ABC is an 16 point scale and ratings should consist of whole numbers (0 to 100) for each item. Total the ratings and divide by 16 to get each subject's ABC score.
Combined Balance assessment | 15 minutes
  Mini Balance Evaluation System Test (mini-BESTest) will be used and it assesses 4 domains: Anticipatory postural adjustments, Reactive postural control, Sensory orientation, and Dynamic gait. The test has a maximum score of 28 points from 14 items that are each scored from 0-2. "0" indicates the lowest level of function and "2" the highest level of function.

OTHER OUTCOMES:
Qualitative Data | 45 minutes
  Interviews with participants and a focus group for research assistants will explore perceived barriers and facilitators, including feasibility, acceptability, usability, and safety, for implementing the assessment. Face-to-face semi-structured interviews for participants will take place at Ain Shams University Hospital, while an online meeting will be arranged for the focus group.

CONTACTS AND LOCATIONS:
Overall Officials: Yasmine S Gomaa, Ph.d, Principal Investigator — Kafrelsheikh University
Locations (1):
- Human Mechatronics Lab, Ain Shams Virtual Hospital, Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gomaa YS, Awad MI, Emara T, Elbokl A, Al-Yahya E, ElMeligie MM. Role of virtual reality in examining the effect of fear of falling (FOF) on postural stability in individuals without and with Parkinson's disease in Egypt: a mixed-methods feasibility study protocol. BMJ Open. 2024 May 1;14(5):e080592. doi: 10.1136/bmjopen-2023-080592. PMID 38692713